CLINICAL TRIAL: NCT04900480
Title: Pilot Project for Direct Access to Physical Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ulla Toft (Other)
Collaborators: Region Hovedstadens Apotek (Other Government)
Responsible Party: Sponsor-Investigator, Ulla Toft, Head of Department, Lecturer Ph.D, MSc Human Nutrition, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Direct Access
Record Dates: First submitted 2020-02-12; First posted 2021-05-25 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Musculoskeletal Diseases
Keywords: Physiotherapy; Public subsidy; Direct access
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Public subsidy to physiotherapy continue as usual (No Intervention): This control arm consists of all physiotherapy clinics with registered provider numbers in two municipalities, where the access and public subsidy to physiotherapy continue as usual.
- Direct access to publicly subsidized physiotherapy (Experimental): This intervention arm consists of all physiotherapy clinics with registered provider numbers in two municipalities, introducing temporary exemption on the legal required general practitioner referral for public subsidy for treatment in general physiotherapy.
  Interventions: Other: Direct access to publicly subsidized physiotherapy

INTERVENTIONS:
Other: Direct access to publicly subsidized physiotherapy — This pilot project introduces temporary exemption on the legal required GP referral for public subsidy for treatment in general physiotherapy.
  Arms: Direct access to publicly subsidized physiotherapy

SUMMARY:
The aim of this pilot study is to evaluate the effect of publicly subsidized physiotherapy for all patients receiving general treatment in physiotherapy clinics with an official provider number. This study will evaluate effects on physical and mental health, number of consultations in physiotherapy; number of contacts with general practitioner; referrals to diagnostic imaging; number of contacts with specialists within rheumatology, neurology and orthopedics and patient satisfaction.

DETAILED DESCRIPTION:
In Denmark, patients in physiotherapy with a referral from their general practitioner (GP) get 40% of their expenses paid by public subsidy. This study aims to test the effects of direct access to physiotherapy with public subsidy without a referral from the GP.

GPs are by default the gatekeeper to all public health care services in Denmark. However, increasing demand in terms of task complexity and patient volume is putting pressure on GPs. In this study, physiotherapists may become the first point of access for patients with musculoskeletal problems.

The hypothesis is, that direct access may decrease use of health services and increase patient satisfaction by shortening the time between occurrence of symptoms and beginning treatment in physiotherapy a) by eliminating the time needed to get a referral from the GP and b) by making access to physiotherapy easier, thus encouraging patients to seek and begin treatment earlier.

The effect of direct access to physiotherapy with public subsidy will be tested in a controlled design. Four similar municipalities located in the Capital Region of Denmark were selected to participate in the study. The four municipalities have been grouped in pairs to ensure similarity on size, health utilization, urbanization and commuting patterns. Two grouped municipalities have been assigned to the intervention group by lottery; the matching pair of municipalities have been assigned to the control group.

From November 2020 to November 2021, citizens living in the two intervention municipalities can get public subsidy for general physiotherapy without a GP referral. For all citizens in the control group access to physiotherapy is provided as usual; thus, public subsidy physiotherapy is only provided for patients with a GP referral. The study includes all physiotherapy clinics in all four municipalities. All included clinics must have an official provider number, i.e. be approved to offer services with public subsidy.

All patients with residence within one of the four municipalities who seeks general treatment in included physiotherapy clinics within their own municipality will be invited to participate in the study. Both patients with and without a GP referral will be included. Participation involves giving consent to providing data for the evaluation.

Data in the study consists of health care contacts accessed through the Capital Region of Denmark's own price mechanism registers logging all transactions between relevant service providers and the Capital Region of Denmark. In addition, all patients are asked to fill in a survey before their 1st diagnostic consultation with a physiotherapist and a follow up survey at six weeks and six months. Finally, the study will collect data through interviews with general practitioners and physiotherapists as well as their respective receptionists.

ELIGIBILITY:
Inclusion Criteria:

* Begin treatment in general physiotherapy within the four municipalities included

Exclusion Criteria:

* Pregnancy
* Have a GP referral to home treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2427 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline physical functioning at 6 months | Six months
  Physical functioning will be measured by a validated Danish Short Form 12 instrument. The questionnaire consists of six items weighted, summed and transformed to provide physical health score. The score of 50 represents the median score of a reference population. 10 points equals 1 standard deviation. Higher score equal better physical health.
Consultations in general practice | Six months after intervention period
  Number of consultations in general practice

SECONDARY OUTCOMES:
Consultations with specialists within rheumatology | Six months after intervention period
  Number of Consultations with specialists within rheumatology
Consultations with specialists within neurology | Six months after intervention period
  Number of consultations with specialists within neurology
Consultations with specialists within orthopedics | Six months after intervention period
  Number of consultations with specialists within orthopedics
Referrals to diagnostic imaging | Six months after intervention period
  Number of referrals to diagnostic imaging
Cancer diagnoses | Five years after intervention period
  Number of cancer diagnoses
Change from baseline physical functioning at six weeks | Six months
  Physical functioning will be measured by a validated Danish Short Form 12 instrument. The questionnaire consists of six items weighted, summed and transformed to provide physical health score. The score of 50 represents the median score of a reference population. 10 points equals 1 standard deviation. Higher score equal better physical health.
Change from baseline mental health at six weeks | Six weeks
  Mental health will be measured by a validated Danish Short Form 12 instrument. The questionnaire consists of six items weighted, summed and transformed to provide mental health score. The score of 50 represents the median score of a reference population. 10 points equals 1 standard deviation. Higher score equal better mental health.
Change from baseline mental health at six months | Six months
  Mental health will be measured by a validated Danish Short Form 12 instrument. The questionnaire consists of six items weighted, summed and transformed to provide mental health score. The score of 50 represents the median score of a reference population. 10 points equals 1 standard deviation. Higher score equal better mental health.
Change from baseline pain intensity at 6 months | Six months
  Pain intensity will be measured by Numeric Rating Scale. The score ranges from 0-10, with 0 indicating no pain and 10 worst possible pain.
Patient satisfaction | Six weeks
  Patient satisfaction will be measured by an overall satisfaction question with five levels of severity. Answers will be scored from 1-5.
  1 = lowest satisfaction, 5 = highest satisfaction.
Patient satisfaction | Six months
  Patient satisfaction will be measured by an overall satisfaction question with five levels of severity. Answers will be scored from 1-5.
  1 = lowest satisfaction, 5 = highest satisfaction.
Trust in collaboration between physiotherapist and general practitioner | Six months
  Patient perceived trust in professional collaboration between physiotherapist and general practitioner will be measured by questionnaire consisting of three questions with 5 levels of severity. Answers will be scored from 1-5.
  1 = lowest satisfaction, 5 = highest satisfaction.
Change in sickness absence | Six weeks
  Sickness absence is measured by two questionnaire items indicating number of full sickness absence days and number of partial sickness absence days the last 30 days. Answers will be between 0-30 for both questions. Fewer days of sickness absence is a better outcome.
Change in sickness absence | Six months
  Sickness absence is measured by two questionnaire items indicating number of full sickness absence days and number of partial sickness absence days the last 30 days. Answers will be between 0-30 for both questions. Fewer days of sickness absence is a better outcome.
Change in use of pharmaceuticals | Six weeks
  Use of pharmaceuticals is measured by two questionnaire items indicating number of days of using over the counter painkillers and number og days using prescribed painkillers on average the last three months. The questions have four levels of severity (0, 1-7, 8-15, 16-30 days on average the last three months). Use of less pharmaceuticals is a better outcome.
Change in use of pharmaceuticals | Six months
  Use of pharmaceuticals is measured by two questionnaire items indicating number of days of using over the counter painkillers and number og days using prescribed painkillers on average the last three months. The questions have four levels of severity (0, 1-7, 8-15, 16-30 days on average the last three months). Use of less pharmaceuticals is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Toft, ph.d., Study Director — Center for Clinical Research and Prevention
Locations (1):
- Center for Clinical Research and Prevention, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahlerup J, Toft U, Schiotz ML, Grew J, Thrysoe R, Ottosen J, Jakobsen LM. Protocol for a cluster-randomized non-inferiority trial of the effect of direct access to publicly subsidized physiotherapy for adults with musculoskeletal pain. Contemp Clin Trials. 2022 Feb;113:106648. doi: 10.1016/j.cct.2021.106648. Epub 2021 Dec 10. PMID 34896641